CLINICAL TRIAL: NCT04408261
Title: Buqitongluo Granule for Qi Deficiency and Blood Stasis Syndrome: A Multicenter, Randomized, Double-blind, Placebo-Controlled Trial
Brief Title: BuqitongluO Granule for Qi Deficiency and Blood Stasis Syndrome
Acronym: BOSS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Collaborators: The Affiliated Hospital of Changchun University of Chinese Medicine (Unknown); The Affiliated Hospital of Shandong University of Chinese Medicine (Unknown); Chengdu University of Traditional Chinese Medicine (Other); The Second Affiliated Hospital of Tianjin University of Traditional Chinese Medicine (Unknown); First Affiliated Hospital of Heilongjiang Chinese Medicine University (Other); Second Affiliated Hospital of Heilongjiang University of Chinese Medicine (Other); The Second Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other); Hunan Academy of Traditional Chinese Medicine Affiliated Hospital (Unknown); The First Clinical Hospital of Jilin Academy of Traditional Chinese Medicine (Unknown); Shaanxi Buchang Pharmaceuticals Co., Ltd. (Unknown); Beijing Chuanglikechuang Medical Technology Development Co., Ltd. (Unknown); Shanghai Youningwei Biotechnology Co., Ltd. (Unknown); Wuhan Zhizhi Medical Technology Co., Ltd. (Unknown); Wuhan Third Hospital (Other); Rizhao Hospital of Traditional Chinese Medicine (Unknown); The First Affiliated Hospital of Guangxi University of Traditional Chinese Medicine (Unknown); Jiangbin Hospital of Guangxi Zhuang Autonomous Region (Unknown)
Responsible Party: Principal Investigator, Ying Gao, President of the Institute for Brain Disorders, Beijing University of Chinese Medicine, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017L04609
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2020-05

CONDITIONS: Stroke, Ischemic; Coronary Artery Disease; Angina Pectoris, Stable; Diabetic Peripheral Neuropathy
Keywords: Qi Deficiency and Blood Stasis Syndrome; Buqitongluo Granule; Traditional Chinese Medicine; Double-Blind; Randomized Controlled Trial
MeSH Terms: conditions — Ischemic Stroke; Coronary Artery Disease; Angina, Stable | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buqitongluo Granule (Experimental): Subjects will receive orally administered Buqitongluo Granules, combined with guidelines-based standard care.
  Interventions: Drug: Buqitongluo Granule; Other: Standard care
- Placebo (Placebo Comparator): Subjects will receive orally administered Buqitongluo Granule placeboes, combined with guidelines-based standard care.
  Interventions: Drug: Buqitongluo Granule Placebo; Other: Standard care

INTERVENTIONS:
Drug: Buqitongluo Granule — Buqitongluo Granules were dissolved with boiled water, administered orally, each bag of 10 grams, one bag each time, three times a day for 42 days.
  Arms: Buqitongluo Granule
Drug: Buqitongluo Granule Placebo — Buqitongluo Granule placeboes were dissolved with boiled water, administered orally, each bag of 10 grams, one bag each time, three times a day for 42 days.
  Arms: Placebo
Other: Standard care — Guidelines-based standard care for convalescence of ischemic stroke, stable angina pectoris of coronary artery disease or diabetic peripheral neuropathy.

SUMMARY:
The main purpose of this trial is to evaluate the efficacy and safety of Buqitongluo Granule in treating qi deficiency and blood stasis syndrome, and explore the effect of the improvement of qi deficiency and blood stasis syndrome on the prognosis of diseases.

DETAILED DESCRIPTION:
The BOSS study is a multicenter, randomized, double-blind, placebo-controlled clinical trial. The primary hypothesis of this trial is that Buqitongluo Granule will improve the syndrome score of Qi Deficiency and Blood Stasis in convalescence of ischemic stroke, stable angina pectoris of coronary artery disease and diabetic peripheral neuropathy with qi deficiency and blood stasis syndrome. Buqitongluo Granule will be compared to placebo, combined with guidelines-based standard care in patients. During the trial, it is forbidden to use acupuncture, Traditional Chinese Medicine decoction (compound granule), Traditional Chinese Medicine injection, Chinese patent medicine (including external use), external washing of Traditional Chinese Medicine and health product (composition or efficacy similar to the study drug).

ELIGIBILITY:
Convalescence of ischemic stroke

Inclusion Criteria:

* Diagnosis of qi deficiency and blood stasis syndrome
* Diagnosis of ischemic stroke
* Age ≥ 35 and ≤ 80 years
* The interval from the onset to recruitment was 14-30 days
* NIHSS score ≥ 4 and ≤ 22
* Patient or legally authorized representative has signed informed consent.

Exclusion Criteria:

* Confirmed secondary stroke caused by tumor, brain trauma, or hematological diseases by clinical examination;
* Other conditions that lead to motor dysfunction (e.g. lameness, osteoarthrosis, rheumatoid arthritis, gouty arthritis), which render the neurological function examination unlikely to be assessed;
* Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg), or renal or hepatic insufficiency (hepatic insufficiency is defined as an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value that is 1.5 times the upper limit of normal, renal insufficiency is defined as a serum creatinine concentration value that is over the upper limit of normal);
* Other conditions or mental disorders which according to the judgement of researchers that restrict evaluation of mental function or render outcomes or follow-up unlikely to be assessed;
* Woman with pregnancy, lactation, or woman who wants to be pregnant in recent;
* Patient who is allergic to the study drug or has severe allergic constitution;
* Patient with yellow thick slimy tongue coating;
* Patient who has been participated in other drug or device clinical trials in recent 3 months.

Stable angina pectoris of coronary artery disease

Inclusion Criteria:

* Diagnosis of qi deficiency and blood stasis syndrome
* Diagnosis of stable angina pectoris of coronary artery disease
* Age ≥ 35 and ≤ 80 years
* Canadian Cardiovascular Society (CCS) Classification of Angina Pectoris classⅠ-Ⅲ
* Patient or legally authorized representative has signed informed consent.

Exclusion Criteria:

* Acute coronary syndrome or unstable angina pectoris in the prior 3 months, or other heart diseases (e.g. cardiomyopathy, pericardial disease);
* Severe cardiopulmonary insufficiency (congestive heart failure NYHA class IV, severe abnormal pulmonary function), or severe arrhythmias (e.g. rapid atrial fibrillation, atrial flutter, paroxysmal ventricular tachycardia);
* Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg), or renal or hepatic insufficiency (hepatic insufficiency is defined as an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value that is 1.5 times the upper limit of normal, renal insufficiency is defined as a serum creatinine concentration value that is over the upper limit of normal);
* Other conditions or mental disorders which according to the judgement of researchers that restrict evaluation of mental function or render outcomes or follow-up unlikely to be assessed;
* Woman with pregnancy, lactation, or woman who wants to be pregnant in recent;
* Patient who is allergic to the study drug or has severe allergic constitution;
* Patient with yellow thick slimy tongue coating;
* Patient who has been participated in other drug or device clinical trials in recent 3 months.

Diabetic peripheral neuropathy

Inclusion Criteria:

* Diagnosis of qi deficiency and blood stasis syndrome
* Diagnosis of diabetic peripheral neuropathies
* Age ≥ 35 and ≤ 80 years
* Patient or legally authorized representative has signed informed consent.

Exclusion Criteria:

* HbA1c >10% in the screening period;
* Acute critical disease of diabetes mellitus in the prior 3 months (e.g. hyperglycemia and hypertonic syndrome, diabetic lactic acidosis, diabetic ketoacidosis);
* Severe heart disease, brain disease, or kidney disease;
* Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg), or renal or hepatic insufficiency (hepatic insufficiency is defined as an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value that is 1.5 times the upper limit of normal, renal insufficiency is defined as a serum creatinine concentration value that is over the upper limit of normal);
* Patient with spinal cord injury, cervical or lumbar vertebra disease (nerve root compression, spinal stenosis, cervical or lumbar vertebra degenerative disease), or sequelae of cerebrovascular disease, neuromuscular junction or muscular disease;
* Neuropathies caused by other diseases (e.g. Guillain-Barre syndrome, chronic inflammatory demyelinating polyneuropathy (CIDP), VitB deficiency, hypothyroidism, alcoholism, severe arteriovenous vasculopathy such as venous embolism, lymphangitis);
* Other conditions or mental disorders which according to the judgement of researchers that restrict evaluation of mental function or render outcomes or follow-up unlikely to be assessed;
* Woman with pregnancy, lactation, or woman who wants to be pregnant in recent;
* Patient who is allergic to the study drug or has severe allergic constitution;
* Patient with yellow thick slimy tongue coating;
* Patient with red tongue and scanty tongue coating;
* Patient who has been participated in other drug or device clinical trials in recent 3 months.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in the syndrome score of Qi Deficiency and Blood Stasis | Baseline, at day 14, day 28, day 42 during treatment, and at day 14 after treatment
  The dynamic evaluation will be defined by Evaluation Scale of Qi Deficiency and Blood Stasis Syndrome. The Evaluation Scale of Qi Deficiency and Blood Stasis Syndrome score ranges from 0 (best score) to 51 (worst score).

SECONDARY OUTCOMES:
Neurological impairment will be evaluated by National Institute of Health Stroke Scale (NIHSS) for convalescence of ischemic stroke | Baseline, at day 14, day 28, day 42 during treatment
  The NIHSS score ranges from 0 (best score) to 42 (worst score).
Self-rating symptoms will be evaluated by Visual Analog Scale (VAS) for convalescence of ischemic stroke | Baseline, at day 14, day 28, day 42 during treatment, and at day 14 after treatment
  Including limb numbness, swelling of hands or feet, spontaneous sweating (hemilateral sweating). Participants rated their symptoms on the 100 millimeter (mm) Visual Analog Scale (VAS) ranging from 0 mm (no symptom) to 100 mm (worst symptom).
Continuous changes of Modified Rankin Scale for convalescence of ischemic stroke | Baseline, at day 42 during treatment, and at 90 days after onset
  The Modified Rankin Scale score ranges from 0 (best score) to 6 (worst score).
Activities of daily living will be measured by Barthel Index (BI) score for convalescence of ischemic stroke | Baseline, at day 42 during treatment, and at 90 days after onset
  The Barthel Index score ranges from 0 (worst score) to 100 (best score).
Quality of life will be measured by Short Form 36 (SF-36) Quality of Life Scale for convalescence of ischemic stroke | Baseline, at day 42 during treatment, and at 90 days after onset
  The SF-36 quality of life scale is used to monitor change in subject reported functionality, well-being, and overall health status. The score of each part ranges from 0 (worst score) to 100 (best score).
Change of the Seattle Angina Questionnaire (SAQ) Score for stable angina pectoris of coronary artery disease | Baseline, at day 28 during treatment, at day 14 after treatment, and at 90 days after recruitment
  The maximum score is 100, and the higher the score, the better the quality of life and the state of body function of patient.
Self-rating symptoms will be evaluated by Visual Analog Scale (VAS) for stable angina pectoris of coronary artery disease | Baseline, at day 14, day 28, day 42 during treatment, and at day 14 after treatment
  Including chest tightness, chest pain, palpitation, fatigue, spontaneous sweating. Participants rated their symptoms on the 100 millimeter (mm) Visual Analog Scale (VAS) ranging from 0 mm (no symptom) to 100 mm (worst symptom).
Change of the Clinical Scoring System of Toronto (TCSS) for diabetic peripheral neuropathy | Baseline, at day 14, day 28, day 42 during treatment, at day 14 after treatment, and at 90 days after recruitment
  TCSS includes a score of neural symptoms, nerve reflex scores and sensory examination. The TCSS score ranges from 0 (best score) to 19 (worst score).
Self-rating symptoms will be evaluated by Visual Analog Scale (VAS) for diabetic peripheral neuropathy | Baseline, at day 14, day 28, day 42 during treatment, and at day 14 after treatment
  Including local pain, limb numbness, paresthesia (e.g. burning sensation, formication, electrical sensation). Participants rated their symptoms on the 100 millimeter (mm) Visual Analog Scale (VAS) ranging from 0 mm (no symptom) to 100 mm (worst symptom).
Quality of life will be measured by Short Form 36 (SF-36) Quality of Life Scale for stable angina pectoris of coronary artery disease and diabetic peripheral neuropathy | Baseline, at day 42 during treatment, and at 90 days after recruitment
  The SF-36 quality of life scale is used to monitor change in subject reported functionality, well-being, and overall health status. The score of each part ranges from 0 (worst score) to 100 (best score).

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, MD, Principal Investigator — Dongzhimen Hospital
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu W, Zhou L, Feng L, Zhang D, Zhang C, Gao Y; behalf of the BOSS Group. BuqiTongluo Granule for Ischemic Stroke, Stable Angina Pectoris, Diabetic Peripheral Neuropathy with Qi Deficiency and Blood Stasis Syndrome: Rationale and Novel Basket Design. Front Pharmacol. 2021 Oct 18;12:764669. doi: 10.3389/fphar.2021.764669. eCollection 2021. PMID 34733163